CLINICAL TRIAL: NCT06911567
Title: An Open-Label, Randomized, Crossover Study to Assess the Comparative Bioavailability of New TEV-56286 Formulations Compared to a Reference TEV-56286 Capsule Formulation Following Single-Dose Administration in Healthy Participants
Brief Title: A Study to Assess New Formulations of TEV-56286
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TV56286-BA-10218
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Random sequence of test and reference formulations
  Interventions: Drug: TEV-56286 Test; Drug: TEV-56286 Reference
- Cohort 2 (Experimental): Random sequence of test and reference formulations
  Interventions: Drug: TEV-56286 Test; Drug: TEV-56286 Reference

INTERVENTIONS:
Drug: TEV-56286 Test — Administered orally
  Other Names: Emrusolmin
Drug: TEV-56286 Reference — Administered orally
  Other Names: Emrusolmin

SUMMARY:
The primary objective of the study is to assess the relative bioavailability of TEV-56286 test formulations compared to TEV-56286 reference product in healthy adult participants.

The secondary objective is to evaluate the safety and tolerability of TEV-56286.

The planned duration for each participant is approximately 70 days which includes a 45 day screening period.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 kg/m2 to 32.0 kg/m2 (inclusive)
* Females of childbearing potential agree to take appropriate measures to prevent pregnancy during the study
* Males who do not have a documented vasectomy or are not congenitally sterile must agree to abstinence or use of barrier method with spermicide with female partner. Male participant who is having sexual intercourse with a woman of childbearing potential who is not currently pregnant will be advised of her requirement to use an additional highly effective contraceptive method
* NOTE - Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Participation in another clinical trial simultaneously
* Females who are lactating, breastfeeding, or intends to become pregnant over the course of the study
* History of alcohol, drug or any other substance, abuse, addiction or dependence in the last 12 months (except for caffeine)
* Major trauma or surgery in the 2 months before screening or at any time between screening and the first dose of IMP, or surgery scheduled during the study or follow-up period
* Donated blood or blood products (eg, white blood cells [WBCs], platelets, etc.) within the 60 days before screening, or has donated blood or blood products at least twice within the 6 months before screening, or has donated plasma within 7 days of the screening visit or has received blood or blood products in the 6 weeks before screening
* Personal or family history of arrhythmia, sudden unexplained death at a young age (before 40 years) in a first-degree relative, or long QT syndrome, or a personal history of syncope, or previous personal treatment for high blood pressure
* NOTE - Additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Drug Concentration (Cmax) | Up to Day 17
Area Under the Drug Concentration-Time Curve from Time 0 to Last Measurable Drug Concentration [AUC(0-t)] | Up to Day 17
Area Under the Drug Concentration-Time Curve from Time 0 to Infinity [AUC(0-inf)] | Up to Day 17

SECONDARY OUTCOMES:
Number of participants with at least one treatment-emergent adverse event | Up to Day 26
Number of participants who did not complete the trial due to an adverse event | Up to Day 26

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D LLC
Locations (1):
- Teva Investigational Site 12141, Miramar, Florida, United States

IPD SHARING:
Plan to Share IPD: No